CLINICAL TRIAL: NCT04024917
Title: Implementation of a Cardiac Coherence Program to Reduce Anxiety in Patients With Peritoneal Carcinosis Treated by Surgery: Randomized Pilot Study
Brief Title: Impact of Cardiac Coherence on Anxiety in Patients Operated on for a Peritoneal Carcinosis
Acronym: COCOON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2019-12 COC
Record Dates: First submitted 2019-07-15; First posted 2019-07-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Peritoneal Carcinomatosis; Pseudomyxoma Peritonei; Mesothelioma Peritoneum
Keywords: Colon; Rectum; Stomach; Ovary
MeSH Terms: conditions — Peritoneal Neoplasms; Pseudomyxoma Peritonei | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coherence cardiac (Experimental)
  Interventions: Other: Cardiac coherence
- Standard care (Active Comparator)
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Cardiac coherence — An initiation session to cardiac coherence will take place D-11 before the operation (during the surgical consultation) in order to obtain a breathing rate of 6 cycles/min via a free application (Respirelax) with listening to an audio tape.
  3 cardiac coherence sessions per day of 5 min (before meals) during the 11 days preceding the operation.
  - The program cardiac coherence will be performed during 90 days after the surgery
  Arms: Coherence cardiac
Other: Standard care — Standard care
  Arms: Standard care

SUMMARY:
The investigator proposes to use the cardiac coherence technique to diminish anxiety before the surgery of a peritoneal carcinosis of colon or stomach or ovary and pseudomyxoma or peritoneal mesothelioma.

DETAILED DESCRIPTION:
Facing a Peritoneal Carcinomatosis (PC) diagnosis requires significant psychological adjustments that may generate major distress because of heavy care and a sometimes poor prognosis. Psychological distress, which most frequently results in emotional anxiety and depressive disorders, affects nearly 40% of patients in oncology. These disorders impair their quality of life, their health behaviours, their therapeutic alliance with caregivers, and represent a risk factor for mortality since access to care, lifestyle and therapeutic adherence differ. All learned societies (e.g., American Society of Clinical Oncology - ASCO), associations (e.g., Union for International Cancer Control (UICC), World Cancer Research Fund International - WCRF) and authorities (e.g., French National Institute of Cancer) recommend both the screening and treatment of this psychological distress. This complementary therapy should be integrated in the overall management of cancer patients, especially since anxiolytics (e.g., benzodiazepines) have shown limitations in clinical trials compared with placebo or standard care. Studies evaluating relevant psychological interventions to treat these disorders are rare. It is therefore essential to assess the feasibility and relevance of implementing a non-drug intervention known for its anxiolytic and antidepressant effects, to respond early and appropriately to the distress and anxiety of patients with PC before and after their surgery. Among the various existing non-drug interventions, a targeted cardiac coherence program seems promising. Cardiac coherence corresponds to a physiological state of balance of the autonomic nervous system obtained through precise and rigorous breathing exercises. Several pilot studies justify its interest in oncology. The main objective of this study is to evaluate adherence to a cardiac coherence program aimed at reducing anxiety in patients with PC awaiting cytoreductive surgery. The secondary objectives are to evaluate the implementation of this program in a cancer center, its adoption by the patients and the impact of this practice on their anxious symptomatology, immunological response and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Patients with peritoneal carcinosis awaiting cytoreductive surgery
3. Patients who scored strictly above 3 on the visual analogue anxiety scale and/or the psychological distress scale
4. Patients with sufficient command of the French language
5. Patient affiliated to a French social security system
6. Patient hospitalized at the Institute of cancer of Montpellier the day before his cytoreductive surgery (at T1 = D-1)
7. Signing of informed consent before any specific trial procedure

Exclusion Criteria:

1. Patients who already have daily practice of cardiac coherence
2. Presence of proven psychiatric disorders (e.g., mental retardation, psychotic disorders, learning disabilities, attention deficit/hyperactivity, bipolar disorder, etc.) other than mood disorders that are reactive to the disease experience, or receiving psychotic treatment that may impair thinking, judgment or discernment
3. Physical or sensory inability to respond to questionnaires
4. Patients who have had a heart transplant or bypass surgery in the Year before surgery
5. Patient with a history of uncontrolled neurological pathology within the last 6 months before inclusion in the trial
6. Patients with a history of psychoactive substance dependence (excluding smoking) in the last 6 months before inclusion in the trial
7. Patients with brain metastases
8. Known natural bradycardia 50 beats per minute
9. Beta-blocker intake in progress
10. Ongoing cardiac arrhythmias
11. Known severe heart failure with ventricular ejection fraction strictly Below 40 %
12. Chronic uncontrolled pain and making it difficult to practice the technique
13. Patient with chronic obstructive pulmonary disease
14. Legal incapacity (patient under guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac Coherence Program Adherence Rate | Around 10 days
  Cardiac Coherence Program Adherence Rate. Patients are considered in "success" adhere to the program) if they will perform at least 20 of the 30 sessions scheduled until surgery (minimum 1 practice per day).

SECONDARY OUTCOMES:
Anxiety by using the visual analogue scale (VAS) | 90 days
  This scale measures the anxiety of patient. It's a visual analogue scale which is also known as linear analogue scale. These scales require respondents to place a mark on a line on which opposing statements or descriptions are placed at either end of a (usually) 10 cm line. The points at which respondents make their mark represent where they perceive their answer to lie in this continuum. The distance between their mark and one end (or the mid-point) of the scale is recorded. The position on the left being the absence of anxiety and the position on the right an unbearable anxiety.
Anxiety and depression by using the hospital anxiety and depression scale (HADS) | 90 days
  One subscale for evaluation of anxiety from 0 (lower anxiety) to 21 (higher anxiety) and the other subscale for depression from 0 (lower anxiety) to 21 (higher depression)
Psychological distress scale | 90 days
  This scale measures the psychological distress of the patient . Psychological distress is characterized by the presence of symptoms, most often depressive or anxious.It's a visual analogue scale which is also known as linear analogue scale. These scales require respondents to place a mark on a line on which opposing statements or descriptions are placed at either end of a line. The position of the mark on the top is the higher psychological distress and at the bottom the lower psychological distress.
Generalized anxiety by using Freeston's uncertainty tolerance scale | 90 days
  The scale is used to identify people with generalized anxiety disorder compared to people with other anxiety disorders or people without pathologies. Range is from 27 (lower uncertainty) to 135 (higher uncertainty)
Heart rate variability | 90 days
  The heart rate variability is determined by using the software EmWave Pro which measures the ratio low frequencies/high frequencies.
Quality of life by using the quality of life questionnaire score (QLQ-C30) | 90 days
  The EORTC QLQ-C30 uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Number of days of hospitalization after surgery | 1 month
Pain by using the visual analogue scale (VAS) | 90 days
  This scale measures the pain of patient. It's a visual analogue scale which is also known as linear analogue scale. These scales require respondents to place a mark on a line on which opposing statements or descriptions are placed at either end of a (usually) 10 cm line. The points at which respondents make their mark represent where they perceive their answer to lie in this continuum. The distance between their mark and one end (or the mid-point) of the scale is recorded. The position on the left being the absence of pain and the position on the right an unbearable pain.
Concentration of salivary immunoglobulin A | 90 days
Number of cardiac coherence sessions per day and by patient | Through the study, an average of 1 year
Reasons of non-participation reported by patients and registered in the form of inclusion | Through study completion, an average of 1 year
Number of patients satisfied with the cardiac coherence program | 90 days
Subjective anxiety score by using the state-trait anxiety inventory form A (STAI-Y form A) questionnaire | 90 days
  State anxiety reflects the current emotional state, which allows the patient's nervousness and worry to be assessed during the session. The range is from 20 (lower anxiety) to 80 (higher anxiety). The patient must answer 20 questions for each part, each answer being on a 4 point Likert scale.
Subjective anxiety score by using the state-trait anxiety inventory form B (STAI-Y form B) questionnaire | 90 days
  Trait anxiety reflects the usual emotional state. The range is from 20 (lower anxiety) to 80 (higher anxiety).The patient must answer 20 questions for each part, each answer being on a 4 point Likert scale
Composite anxiety symptomatology score | 90 days
  Score including psychological, physiological and biological variables
Feedback from the instructor and investigator | 90 days
Recruitment and retention rates | 1 year
Duration of cardiac coherence sessions in minutes | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Estelle Guerdoux-Ninot, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (1):
- ICM, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Yes
All data will be available after publication of the results in peer-reviewed revues, and in national and international meetings. It includes all disidentified participants' data, the study protocol, the statistical analysis plan and analytic code. The corresponding author will provide data and datasets generated and/or analyzed during the study upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Access to study data upon written detailed request sent to ICM, following publication and until 5 years after publication of summary data.
Access Criteria: The data shared will be limited to that required for independent mandated verification of the published results, the applicant will need authorization from ICM for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Dodson RM, McQuellon RP, Mogal HD, Duckworth KE, Russell GB, Votanopoulos KI, Shen P, Levine EA. Quality-of-Life Evaluation After Cytoreductive Surgery with Hyperthermic Intraperitoneal Chemotherapy. Ann Surg Oncol. 2016 Dec;23(Suppl 5):772-783. doi: 10.1245/s10434-016-5547-y. Epub 2016 Sep 8. PMID 27638671
- [Background] Lloyd-Williams M, Dennis M, Taylor F. A prospective study to determine the association between physical symptoms and depression in patients with advanced cancer. Palliat Med. 2004 Sep;18(6):558-63. doi: 10.1191/0269216304pm923oa. PMID 15453627
- [Background] Pinquart M, Duberstein PR. Depression and cancer mortality: a meta-analysis. Psychol Med. 2010 Nov;40(11):1797-810. doi: 10.1017/S0033291709992285. Epub 2010 Jan 20. PMID 20085667
- [Background] Elkins G, Staniunas R, Rajab MH, Marcus J, Snyder T. Use of a numeric visual analog anxiety scale among patients undergoing colorectal surgery. Clin Nurs Res. 2004 Aug;13(3):237-44. doi: 10.1177/1054773803262222. PMID 15245638
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Sugarbaker PH. Peritonectomy procedures. Ann Surg. 1995 Jan;221(1):29-42. doi: 10.1097/00000658-199501000-00004. PMID 7826158
- [Background] Tan G, Dao TK, Farmer L, Sutherland RJ, Gevirtz R. Heart rate variability (HRV) and posttraumatic stress disorder (PTSD): a pilot study. Appl Psychophysiol Biofeedback. 2011 Mar;36(1):27-35. doi: 10.1007/s10484-010-9141-y. PMID 20680439
- [Background] Bartos A, Bartos D, Raluca S, Mitre C, Hadade A, Iancu I, Cioltean C, Iancu C, Militaru C, Parau A, Breazu C. Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy for the Treatment of Peritoneal Carcinomatosis: Our Initial Experience. Chirurgia (Bucur). 2019 Mar-Apr;114(2):222-233. doi: 10.21614/chirurgia.114.2.222. PMID 31060655
- [Background] Glehen O, Mohamed F, Sugarbaker PH. Incomplete cytoreduction in 174 patients with peritoneal carcinomatosis from appendiceal malignancy. Ann Surg. 2004 Aug;240(2):278-85. doi: 10.1097/01.sla.0000133183.15705.71. PMID 15273552
- [Background] Piso P, Stierstorfer K, Gerken M, Klinkhammer-Schalke M. Benefit of cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy in patients with isolated peritoneal metastases from colorectal cancer. Int J Colorectal Dis. 2018 Nov;33(11):1559-1567. doi: 10.1007/s00384-018-3146-z. Epub 2018 Aug 21. PMID 30132068
- [Background] Balaphas A, Belfontali V, Ris F, Lanitis A, Meier RP, Amram ML, Roth A, Huber O, Berney T, Morel P. [Management of peritoneal carcinomatosis with cytoreductive surgery and hyperthermic intraperitoneal chemotherapy]. Rev Med Suisse. 2016 Jun 15;12(523):1190-4. French. PMID 27487625
- [Background] Minnella EM, Carli F. Prehabilitation and functional recovery for colorectal cancer patients. Eur J Surg Oncol. 2018 Jul;44(7):919-926. doi: 10.1016/j.ejso.2018.04.016. Epub 2018 Apr 30. PMID 29754828
- [Background] Mitchell AJ, Chan M, Bhatti H, Halton M, Grassi L, Johansen C, Meader N. Prevalence of depression, anxiety, and adjustment disorder in oncological, haematological, and palliative-care settings: a meta-analysis of 94 interview-based studies. Lancet Oncol. 2011 Feb;12(2):160-74. doi: 10.1016/S1470-2045(11)70002-X. Epub 2011 Jan 19. PMID 21251875
- [Background] Carlson LE, Angen M, Cullum J, Goodey E, Koopmans J, Lamont L, MacRae JH, Martin M, Pelletier G, Robinson J, Simpson JS, Speca M, Tillotson L, Bultz BD. High levels of untreated distress and fatigue in cancer patients. Br J Cancer. 2004 Jun 14;90(12):2297-304. doi: 10.1038/sj.bjc.6601887. PMID 15162149
- [Background] Mehnert A, Hartung TJ, Friedrich M, Vehling S, Brahler E, Harter M, Keller M, Schulz H, Wegscheider K, Weis J, Koch U, Faller H. One in two cancer patients is significantly distressed: Prevalence and indicators of distress. Psychooncology. 2018 Jan;27(1):75-82. doi: 10.1002/pon.4464. Epub 2017 Jun 16. PMID 28568377
- [Background] Basak F, Hasbahceci M, Guner S, Sisik A, Acar A, Yucel M, Kilic A, Bas G. Prediction of anxiety and depression in general surgery inpatients: A prospective cohort study of 200 consecutive patients. Int J Surg. 2015 Nov;23(Pt A):18-22. doi: 10.1016/j.ijsu.2015.09.040. Epub 2015 Sep 16. PMID 26384837
- [Background] Kayhan F, Cicek E, Uguz F, Karababa IF, Kucur R. Mood and anxiety disorders among inpatients of a university hospital in Turkey. Gen Hosp Psychiatry. 2013 Jul-Aug;35(4):417-22. doi: 10.1016/j.genhosppsych.2013.03.004. Epub 2013 Apr 18. PMID 23602607
- [Background] Arrieta O, Angulo LP, Nunez-Valencia C, Dorantes-Gallareta Y, Macedo EO, Martinez-Lopez D, Alvarado S, Corona-Cruz JF, Onate-Ocana LF. Association of depression and anxiety on quality of life, treatment adherence, and prognosis in patients with advanced non-small cell lung cancer. Ann Surg Oncol. 2013 Jun;20(6):1941-8. doi: 10.1245/s10434-012-2793-5. Epub 2012 Dec 22. PMID 23263699
- [Background] Foster C, Haviland J, Winter J, Grimmett C, Chivers Seymour K, Batehup L, Calman L, Corner J, Din A, Fenlon D, May CM, Richardson A, Smith PW; Members of the Study Advisory Committee. Pre-Surgery Depression and Confidence to Manage Problems Predict Recovery Trajectories of Health and Wellbeing in the First Two Years following Colorectal Cancer: Results from the CREW Cohort Study. PLoS One. 2016 May 12;11(5):e0155434. doi: 10.1371/journal.pone.0155434. eCollection 2016. PMID 27171174
- [Background] Fox JP, Philip EJ, Gross CP, Desai RA, Killelea B, Desai MM. Associations between mental health and surgical outcomes among women undergoing mastectomy for cancer. Breast J. 2013 May-Jun;19(3):276-84. doi: 10.1111/tbj.12096. Epub 2013 Mar 21. PMID 23521554
- [Background] Wada S, Inoguchi H, Sadahiro R, Matsuoka YJ, Uchitomi Y, Sato T, Shimada K, Yoshimoto S, Daiko H, Shimizu K. Preoperative Anxiety as a Predictor of Delirium in Cancer Patients: A Prospective Observational Cohort Study. World J Surg. 2019 Jan;43(1):134-142. doi: 10.1007/s00268-018-4761-0. PMID 30128769
- [Background] Jamison RN, Parris WC, Maxson WS. Psychological factors influencing recovery from outpatient surgery. Behav Res Ther. 1987;25(1):31-7. doi: 10.1016/0005-7967(87)90112-4. No abstract available. PMID 2954531
- [Background] Prieto JM, Blanch J, Atala J, Carreras E, Rovira M, Cirera E, Gasto C. Psychiatric morbidity and impact on hospital length of stay among hematologic cancer patients receiving stem-cell transplantation. J Clin Oncol. 2002 Apr 1;20(7):1907-17. doi: 10.1200/JCO.2002.07.101. PMID 11919251
- [Background] Scott LE, Clum GA, Peoples JB. Preoperative predictors of postoperative pain. Pain. 1983 Mar;15(3):283-93. doi: 10.1016/0304-3959(83)90063-5. PMID 6856324
- [Background] Kim Y, Spillers RL. Quality of life of family caregivers at 2 years after a relative's cancer diagnosis. Psychooncology. 2010 Apr;19(4):431-40. doi: 10.1002/pon.1576. PMID 19399773
- [Background] Satin JR, Linden W, Phillips MJ. Depression as a predictor of disease progression and mortality in cancer patients: a meta-analysis. Cancer. 2009 Nov 15;115(22):5349-61. doi: 10.1002/cncr.24561. PMID 19753617
- [Background] Cossu G, Saba L, Minerba L, Mascalchi M. Colorectal Cancer Screening: The Role of Psychological, Social and Background Factors in Decision-making Process. Clin Pract Epidemiol Ment Health. 2018 Mar 21;14:63-69. doi: 10.2174/1745017901814010063. eCollection 2018. PMID 29643929
- [Background] Smith SK, Loscalzo M, Mayer C, Rosenstein DL. Best Practices in Oncology Distress Management: Beyond the Screen. Am Soc Clin Oncol Educ Book. 2018 May 23;38:813-821. doi: 10.1200/EDBK_201307. PMID 30231391
- [Background] Wagner LI, Spiegel D, Pearman T. Using the science of psychosocial care to implement the new american college of surgeons commission on cancer distress screening standard. J Natl Compr Canc Netw. 2013 Feb 1;11(2):214-21. doi: 10.6004/jnccn.2013.0028. PMID 23411387
- [Background] Dolbeault S, Boistard B, Meuric J, Copel L, Bredart A. Screening for distress and supportive care needs during the initial phase of the care process: a qualitative description of a clinical pilot experiment in a French cancer center. Psychooncology. 2011 Jun;20(6):585-93. doi: 10.1002/pon.1946. Epub 2011 Mar 22. PMID 21425386
- [Background] Dolbeault S, Bredart A, Mignot V, Hardy P, Gauvain-Piquard A, Mandereau L, Asselain B, Medioni J. Screening for psychological distress in two French cancer centers: feasibility and performance of the adapted distress thermometer. Palliat Support Care. 2008 Jun;6(2):107-17. doi: 10.1017/S1478951508000187. PMID 18501045
- [Background] Maurice-Szamburski A, Auquier P, Viarre-Oreal V, Cuvillon P, Carles M, Ripart J, Honore S, Triglia T, Loundou A, Leone M, Bruder N; PremedX Study Investigators. Effect of sedative premedication on patient experience after general anesthesia: a randomized clinical trial. JAMA. 2015 Mar 3;313(9):916-25. doi: 10.1001/jama.2015.1108. PMID 25734733
- [Background] Karavidas MK, Lehrer PM, Vaschillo E, Vaschillo B, Marin H, Buyske S, Malinovsky I, Radvanski D, Hassett A. Preliminary results of an open label study of heart rate variability biofeedback for the treatment of major depression. Appl Psychophysiol Biofeedback. 2007 Mar;32(1):19-30. doi: 10.1007/s10484-006-9029-z. Epub 2007 Mar 1. PMID 17333315
- [Background] Trousselard M, Canini F, Claverie D, Cungi C, Putois B, Franck N. Cardiac Coherence Training to Reduce Anxiety in Remitted Schizophrenia, a Pilot Study. Appl Psychophysiol Biofeedback. 2016 Mar;41(1):61-9. doi: 10.1007/s10484-015-9312-y. PMID 26346569
- [Background] Berry ME, Chapple IT, Ginsberg JP, Gleichauf KJ, Meyer JA, Nagpal ML. Non-pharmacological Intervention for Chronic Pain in Veterans: A Pilot Study of Heart Rate Variability Biofeedback. Glob Adv Health Med. 2014 Mar;3(2):28-33. doi: 10.7453/gahmj.2013.075. PMID 24808979
- [Background] Haase O, Langelotz C, Scharfenberg M, Schwenk W, Tsilimparis N. Reduction of heart rate variability after colorectal resections. Langenbecks Arch Surg. 2012 Jun;397(5):793-9. doi: 10.1007/s00423-012-0903-2. Epub 2012 Jan 17. PMID 22249435
- [Background] De Couck M, Caers R, Spiegel D, Gidron Y. The Role of the Vagus Nerve in Cancer Prognosis: A Systematic and a Comprehensive Review. J Oncol. 2018 Jul 2;2018:1236787. doi: 10.1155/2018/1236787. eCollection 2018. PMID 30057605
- [Background] Chambers DA. Sharpening our focus on designing for dissemination: Lessons from the SPRINT program and potential next steps for the field. Transl Behav Med. 2020 Dec 31;10(6):1416-1418. doi: 10.1093/tbm/ibz102. PMID 31313812
- [Background] Chambers DA, Norton WE. The Adaptome: Advancing the Science of Intervention Adaptation. Am J Prev Med. 2016 Oct;51(4 Suppl 2):S124-31. doi: 10.1016/j.amepre.2016.05.011. Epub 2016 Jun 28. PMID 27371105
- [Background] Hijazi Y, Gondal U, Aziz O. A systematic review of prehabilitation programs in abdominal cancer surgery. Int J Surg. 2017 Mar;39:156-162. doi: 10.1016/j.ijsu.2017.01.111. Epub 2017 Feb 2. PMID 28161527
- [Background] Abelson JS, Chait A, Shen MJ, Charlson M, Dickerman A, Yeo HL. Sources of distress among patients undergoing surgery for colorectal cancer: a qualitative study. J Surg Res. 2018 Jun;226:140-149. doi: 10.1016/j.jss.2018.01.017. Epub 2018 Feb 22. PMID 29661279
- [Background] Low CA, Bovbjerg DH, Ahrendt S, Alhelo S, Choudry H, Holtzman M, Jones HL, Pingpank JF Jr, Ramalingam L, Zeh HJ 3rd, Zureikat AH, Bartlett DL. Depressive Symptoms in Patients Scheduled for Hyperthermic Intraperitoneal Chemotherapy With Cytoreductive Surgery: Prospective Associations With Morbidity and Mortality. J Clin Oncol. 2016 Apr 10;34(11):1217-22. doi: 10.1200/JCO.2015.62.9683. Epub 2016 Feb 22. PMID 26903574